CLINICAL TRIAL: NCT04607148
Title: A Multicenter, Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of Intravitreal Injections of FHTR2163 in Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: A Study Assessing the Long-Term Safety and Tolerability of Galegenimab (FHTR2163) in Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The benefit to risk balance did not support further treatment with galegenimab (FHTR2163).
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GR42558
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Macular Degeneration, Age-Related; Geographic Atrophy
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will be masked until database lock of the parent study (NCT03972709/GR40973). After the masked period, the study will follow an open-label design. The Outcome Assessor is masked for BCVA assessments.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Galegenimab 20 mg Q4W (Experimental): Participants will receive 20 milligrams (mg) galegenimab via ITV injection every 4 weeks (Q4W).
  Interventions: Drug: Galegenimab
- Galegenimab 20 mg Q8W (Experimental): Participants will receive 20 mg galegenimab via ITV injection every 8 weeks (Q8W).
  Interventions: Drug: Galegenimab
- Galegenimab 10 mg Q4W (Experimental): Participants will receive 10 mg galegenimab via ITV injection Q4W.
  Interventions: Drug: Galegenimab
- Galegenimab 10 mg Q8W (Experimental): Participants will receive 10 mg galegenimab via ITV injection Q8W.
  Interventions: Drug: Galegenimab

INTERVENTIONS:
Drug: Galegenimab — Intravitreal (ITV) injections of galegenimab
  Other Names: FHTR2163

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of intravitreal (ITV) injections of galegenimab (FHTR2163) administered every 4 weeks (Q4W) or every 8 weeks (Q8W) in participants with geographic atrophy (GA) secondary to age-related macular degeneration (AMD) who completed the parent study (NCT03972709/GR40973).

ELIGIBILITY:
Inclusion Criteria:

* Completed the parent study (NCT03972709/GR40973) through the Week 76 visit without early treatment discontinuation
* Sufficiently clear ocular media, adequate pupillary dilation, and fixation to permit acceptable fundus imaging.

Ocular Inclusion Criteria: Study Eye - If the study eye best corrected visual acuity (BCVA) letter score is ≥69 letters (Snellen equivalent of 20/40 or better), the non-study eye must have a BCVA letter score of ≥44 letters (Snellen equivalent of 20/125 or better) on visit Day 1 of the open label extension (OLE)/Week 76 of parent study.

Ocular Inclusion Criteria: Non-Study Eye

- The non-study eye must have a BCVA letter score of ≥44 letters (Snellen equivalent of 20/125 or better) if the study eye BCVA letter score is ≥69 letters (Snellen equivalent of 20/40 or better) on visit Day 1 OLE/Week 76 of parent study.

Exclusion Criteria:

Ocular Exclusion Criteria:

* Active uveitis and/or vitritis (grade trace or above) in either eye
* Active, infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Active or history of choroidal neovascularization (CNV) in study eye that requires anti-vascular endothelial growth factor (anti-VEGF) treatment
* Active or recent history (i.e., since enrollment in parent study) of optic neuritis in either eye
* Retinal pigment epithelium (RPE) tear that involves the macula in either eye
* Moderate or severe non-proliferative diabetic retinopathy in either eye
* Proliferative diabetic retinopathy in either eye
* Central serous retinopathy in either eye
* Recent history of recurrent infectious or inflammatory ocular disease in either eye
* Recent history of idiopathic or autoimmune-associated uveitis in either eye
* Any concurrent ocular or intraocular condition in the study eye that contraindicates the use of an investigational drug or may affect interpretation of the study results or may render the participant at high risk for treatment complications.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (48):
- United States (48):
  - California Retina Consultants, Bakersfield, California
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County, Fullerton, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Consultants, San Diego, Poway, California
  - Retinal Consultants Med Group, Sacramento, California
  - West Coast Retina, San Francisco, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants - Santa Maria, Santa Maria, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Consultants of Southern Colorado PC, Colorado Springs, Colorado
  - Southwest Retina Consultants, Durango, Colorado
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Rand Eye, Deerfield Beach, Florida
  - Florida Eye Associates - Melbourne 2nd Office, Melbourne, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Associates, Tallahassee, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Illinois Eye and Ear Infirmary, Chicago, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Vitreo Retinal Consultants, Wichita, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Associated Retinal Consultants PC, Royal Oak, Michigan
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - NJ Retina Teaneck Clinic, Toms River, New Jersey
  - NJ Retina-Toms River, Toms River, New Jersey
  - Ophthalmic Consultants of Long Island, Oceanside, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates PA, Charlotte, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Cleveland Clinic Foundation; Cole Eye Institute, Cleveland, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Mid Atlantic Retina - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates Chattanooga, Chattanooga, Tennessee
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Spokane Eye Clinical Research, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Galegenimab 10MG Q4W: Participants will receive 10 milligrams (mg) galegenimab via intravitreal (ITV) injection every 4 weeks (Q4W).
- Galegenimab 20MG Q4W: Participants will receive 20 mg galegenimab via ITV injection Q4W.
- Galegenimab 10MG Q8W: Participants will receive 10 mg galegenimab via ITV injection Q8W.
- Galegenimab 20MG Q8W: Participants will receive 20 mg galegenimab via ITV injection Q8W.
Period: Overall Study
Arm/Group | Galegenimab 10MG Q4W | Galegenimab 20MG Q4W | Galegenimab 10MG Q8W | Galegenimab 20MG Q8W
Started | 14 | 70 | 12 | 48
Completed | 0 | 0 | 0 | 0
Not Completed | 14 | 70 | 12 | 48
Not completed — Withdrawal by Subject | 0 | 4 | 2 | 8
Not completed — Study Terminated by Sponsor | 14 | 59 | 9 | 39
Not completed — Sponsor Decision | 0 | 0 | 1 | 0
Not completed — Non-Compliance With Study Drug | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Death | 0 | 3 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galegenimab 10MG Q4W | Galegenimab 20MG Q4W | Galegenimab 10MG Q8W | Galegenimab 20MG Q8W | Total
Number analyzed (Participants) | 14 | 70 | 12 | 48 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.3 (5.4) | 80.2 (7.2) | 78.1 (6.9) | 78.8 (8.5) | 79.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 41 | 6 | 30 | 86
  Male | 5 | 29 | 6 | 18 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 1 | 4
  Not Hispanic or Latino | 14 | 67 | 12 | 47 | 140
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 14 | 69 | 12 | 48 | 143
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Ocular Adverse Events
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition, or any deterioration in a laboratory value or other clinical test. Ocular AEs are the events which are localized in the ocular region.
Time Frame: From baseline up to Week 104
Population: Safety analysis population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Galegenimab 10MG Q4W | Galegenimab 20MG Q4W | Galegenimab 10MG Q8W | Galegenimab 20MG Q8W
Number analyzed (Participants) | 14 | 70 | 12 | 48
Percentage of Participants | 50 | 42.9 | 25 | 27.1

2. Primary Outcome: Percentage of Participants With Systemic (Non-Ocular) Adverse Events
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition, or any deterioration in a laboratory value or other clinical test.
Time Frame: From Baseline up to Week 104
Population: Safety analysis population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Galegenimab 10MG Q4W | Galegenimab 20MG Q4W | Galegenimab 10MG Q8W | Galegenimab 20MG Q8W
Number analyzed (Participants) | 14 | 70 | 12 | 48
Percentage of Participants | 71.4 | 70 | 33.3 | 47.9

ADVERSE EVENTS:
Time Frame: From baseline up to Week 104
Description: Safety analysis population included all randomized participants who received at least one dose of study drug.
Arm/Group | Galegenimab 10MG Q4W | Galegenimab 20MG Q4W | Galegenimab 10MG Q8W | Galegenimab 20MG Q8W
All-Cause Mortality (participants affected / at risk) | 0/14 | 3/70 | 0/12 | 1/48
Serious Adverse Events (participants affected / at risk) | 1/14 | 13/70 | 2/12 | 10/48
Other Adverse Events (participants affected / at risk) | 13/14 | 26/70 | 6/12 | 14/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galegenimab 10MG Q4W (N=14) | Galegenimab 20MG Q4W (N=70) | Galegenimab 10MG Q8W (N=12) | Galegenimab 20MG Q8W (N=48)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Blindness cortical (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal artery spasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastric operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galegenimab 10MG Q4W (N=14) | Galegenimab 20MG Q4W (N=70) | Galegenimab 10MG Q8W (N=12) | Galegenimab 20MG Q8W (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 6 (7) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 2 (2) | 2 (2) | 1 (2) | 2 (2)
Visual impairment (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 3 (3) | 4 (6) | 0 (0) | 0 (0)
Vitritis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 8 (8) | 1 (1) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal foot infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT04607148/Prot_SAP_000.pdf